CLINICAL TRIAL: NCT04521374
Title: Investigating the Influence of Texture Modified and Protein-enriched Meals on Dietary Intake and Appetite Responses in Healthy Older Adults
Brief Title: The Effects of Texture Modified Diets on Dietary Intake and Appetite Responses in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Lisa Methven, : Professor in Food and Sensory Science, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: UREC 19/68
Record Dates: First submitted 2020-08-07; First posted 2020-08-20 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Older Adults
Keywords: Older adults; Texture modified diet; Protein fortification; Appetite; Dietary intake; Food first
MeSH Terms: interventions — Proteins

STUDY DESIGN:
Who Masked: Participant
Masking Description: All samples provided to the participant are labelled with 3 digit random codes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard Meal (Experimental): A regular meal (equivalent to International Dysphagia Diet Standardisation Initiative [IDSSI] Level 7) will consist of meat, potatoes and peas: 333kcal, 16g protein.
  Interventions: Behavioral: Preload meals that are solid or texture modified and are fortified with protein or not fortified with protein
- Standard Protein Fortified Meal (Experimental): A regular meal (equivalent to International Dysphagia Diet Standardisation Initiative [IDSSI] Level 7) will consist of meat, potatoes and peas: 333kcal, 25g protein.
  Interventions: Behavioral: Preload meals that are solid or texture modified and are fortified with protein or not fortified with protein
- Texture Modified Meal (Experimental): A pureed meal (equivalent to International Dysphagia Diet Standardisation Initiative [IDSSI] Level 4) will consist of meat, potatoes and peas: 340kcal, 16g protein.
  Interventions: Behavioral: Preload meals that are solid or texture modified and are fortified with protein or not fortified with protein
- Texture Modified Protein Fortified Meal (Experimental): A pureed meal (equivalent to International Dysphagia Diet Standardisation Initiative [IDSSI] Level 4) will consist of meat, potatoes and peas: 350kcal, 25g protein.
  Interventions: Behavioral: Preload meals that are solid or texture modified and are fortified with protein or not fortified with protein

INTERVENTIONS:
Behavioral: Preload meals that are solid or texture modified and are fortified with protein or not fortified with protein — Immediately after consuming the preload meal, volunteers will use a 100mm visual analogue scale (VAS) to rate their liking towards the meal, their hunger, fullness, desire to eat and prospective food intake. Subsequently, they will record these every 30 minutes until they consume their ad-libitum dinner

SUMMARY:
This study aims to investigate the effects of equicaloric texture modified and regular meals that are either fortified with protein or not on dietary intake and satiety in older adults (65+) living in the United Kingdom (UK).

DETAILED DESCRIPTION:
* To investigate whether there are any differences in appetite responses following a texture modified meal compared to a standard meal.
* To investigate whether protein-enriched versions of a texture modified meal and/or standard meal affects satiety and subsequent intake in healthy older adults.
* To investigate the effects of a texture modified diet, standard diet and their protein-enriched versions on gastric emptying in healthy older adults.

ELIGIBILITY:
Inclusion Criteria:

* aged 65 years or over (no upper age limit);
* be within body mass index range (18.5-34.9kg/m2 );
* regularly consume 3 meals a day (breakfast by 11am, lunch and dinner);
* be able to accept test meals provided;
* be able to feed themselves;
* be able to give informed consent; i.e not lacking mental capacity;
* Have access to a kitchen, freezer and fridge.
* Have access to a telephone.
* understand English.

Exclusion Criteria:

* Diagnosed with coronavirus (COVID-19) or have had it in the last 4 weeks.
* have any existing neurological or gastrointestinal condition;
* have Cancer;
* have no current chewing or swallowing difficulties (such as dysphagia);
* have no existing cognitive or psychiatric disorder;
* taking medications that can significantly affect taste changes, appetite or gastric emptying;
* be on a special or therapeutic diet;
* have any food allergies or intolerances that will be worsened with meals provided in the study;
* have a history of drug or alcohol misuse;
* smoke more than 10 cigarettes a day.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-09-06 (Actual)

PRIMARY OUTCOMES:
Intake at ad-libitum dinner | 4 days in total (one measurement per study day)
  Intake at the ad-libitum meal is measured (grams). Volunteers are instructed to eat only until they feel comfortable satisfied and are given 20 min to consume the meal.

SECONDARY OUTCOMES:
Ratings (Appetite, hedonic and palatability) of breakfast, preload lunch and ad-libitum dinner | Regular ratings each study visit, 4 days in total
  Appetite, hedonic and palatability ratings are assessed using validated 100 mm Visual Analogue Scales (VAS, sscale 0-100). Before and immediately after breakfast and assessed every 30 min for 360 min
Gastric emptying | Regular samples each study visit, 4 days in total
  Gastric emptying will be measured using 13C-labelled sodium acetate which will be added into a bottle of water. This will be consumed alongside preload meal. Measurements will be taken every 1 hour after consumption of breakfast up to preload, then every 15 min after the preload for 180 min.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Methven, BSc, PhD, Principal Investigator — University of Reading
Locations (1):
- University of Reading, Reading, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No personal identification data will be shared. The study is not under an obligation to share data, however, it is possible that some of the individual (unliked / non identifiable) data will be useful in a meta-analysis and, hence sharing individual participant data (IPD) will be considered.

REFERENCES:
- [Background] Wright L, Cotter D, Hickson M, Frost G. Comparison of energy and protein intakes of older people consuming a texture modified diet with a normal hospital diet. J Hum Nutr Diet. 2005 Jun;18(3):213-9. doi: 10.1111/j.1365-277X.2005.00605.x. PMID 15882384
- [Background] Pritchard SJ, Davidson I, Jones J, Bannerman E. A randomised trial of the impact of energy density and texture of a meal on food and energy intake, satiation, satiety, appetite and palatability responses in healthy adults. Clin Nutr. 2014 Oct;33(5):768-75. doi: 10.1016/j.clnu.2013.10.014. Epub 2013 Oct 25. PMID 24200201
- [Background] Keller H, Chambers L, Niezgoda H, Duizer L. Issues associated with the use of modified texture foods. J Nutr Health Aging. 2012 Mar;16(3):195-200. doi: 10.1007/s12603-011-0160-z. PMID 22456772
- [Background] Volkert D, Beck AM, Cederholm T, Cruz-Jentoft A, Goisser S, Hooper L, Kiesswetter E, Maggio M, Raynaud-Simon A, Sieber CC, Sobotka L, van Asselt D, Wirth R, Bischoff SC. ESPEN guideline on clinical nutrition and hydration in geriatrics. Clin Nutr. 2019 Feb;38(1):10-47. doi: 10.1016/j.clnu.2018.05.024. Epub 2018 Jun 18. PMID 30005900
- [Background] Cichero JAY. Age-Related Changes to Eating and Swallowing Impact Frailty: Aspiration, Choking Risk, Modified Food Texture and Autonomy of Choice. Geriatrics (Basel). 2018 Oct 12;3(4):69. doi: 10.3390/geriatrics3040069. PMID 31011104